CLINICAL TRIAL: NCT07195045
Title: Thai Version of PainPREDICT: Translation, Validation, and Mobile Application Development for Screening Painful Diabetic Neuropathy in Diabetes Patients
Brief Title: Thai PainPREDICT Validation Study
Acronym: PainPREDICT-Th
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Jakkrit Amornvit, MD., Priciple Investigator, Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COA No. 1084/2025; IRB No. 0296/68 (Other: Institutional Review Board, Faculty of Medicine, Chulalongkorn University)
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Painful Diabetic Neuropathy (PDN); Diabetic Neuropathy, Distal Symmetric Polyneuropathy (Manifestation); Type 1 Diabetes Mellitus (T1DM); Type 2 Diabetes Mellitus (T2DM); Neuropathic Pain; Diabetes Complications
Keywords: PainPREDICT; Painful Diabetic Neuropathy; Diabetic Neuropathy; Neuropathic Pain Questionnaire; Mobile Health (mHealth); Questionnaire Validation; Screening Tool; Thai Population; Cross-Cultural Adaptation; Digital Health Application; Diabetes Complications; Neuropathy Screening
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Neuralgia; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Participants with type 1 or type 2 diabetes will be divided into two groups: those with painful diabetic neuropathy and those without neuropathy, matched by age, sex, and diabetes type. Both groups will complete the Thai PainPREDICT questionnaire (mobile application and/or paper version). Scores will be compared with clinical diagnosis and neurophysiological testing to assess reliability, validity, and diagnostic accuracy. The model uses parallel assessment rather than crossover or randomized allocation.
Masking Description: Not applicable. Both patients and investigators are aware of PDN status, and the study does not use blinding. Outcomes are assessed by comparing questionnaire/app results with independent clinical and neurophysiological tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Painful Diabetic Neuropathy (PDN) Group (Experimental): Adults with type 1 or type 2 diabetes who have painful diabetic neuropathy, confirmed by clinical assessment. Participants will complete the Thai PainPREDICT questionnaire via the mobile application and/or paper version. Results will be compared against clinical diagnosis and neurophysiological tests.
  Interventions: Diagnostic Test: Thai PainPREDICT Questionnaire and Mobile Application
- Arm 2: Non-PDN Diabetic Control Group (Active Comparator): Adults with type 1 or type 2 diabetes without painful neuropathy, matched by age, sex, and diabetes type. Participants will complete the Thai PainPREDICT questionnaire via the mobile application and/or paper version, with results compared against clinical assessment and neurophysiological testing.
  Interventions: Diagnostic Test: Thai PainPREDICT Questionnaire and Mobile Application

INTERVENTIONS:
Diagnostic Test: Thai PainPREDICT Questionnaire and Mobile Application — The Thai PainPREDICT Questionnaire is a culturally adapted and validated version of an internationally recognized neuropathic pain assessment tool. In this study, it is administered via both paper form and a secure mobile application designed for Thai patients with diabetes. The app automates scoring, provides real-time feedback, and securely stores data in REDCap in compliance with Thai Personal Data Protection Act (PDPA). The intervention is used to screen for painful diabetic neuropathy and compare results against clinical diagnosis and neurophysiological testing, including DN4, nerve conduction studies, and quantitative sensory testing.
  Other Names: PainPREDICT (Thai Version); PainPREDICT App

SUMMARY:
Painful diabetic neuropathy (PDN) is one of the most common and disabling complications of diabetes mellitus, substantially affecting quality of life, daily functioning, and health system burden. Early identification of PDN is crucial for timely treatment, prevention of complications such as foot ulcers and amputations, and for reducing healthcare costs. However, in Thailand there are limited culturally adapted and validated tools for screening PDN. PainPREDICT is an internationally validated questionnaire designed to characterize neuropathic pain profiles, but its adaptation for Thai patients has not yet been undertaken. In parallel, the use of mobile health technologies (mHealth) has the potential to expand access to screening and monitoring of chronic conditions, particularly in resource-limited settings.

DETAILED DESCRIPTION:
This study aims to translate, culturally adapt, and validate the PainPREDICT questionnaire for the Thai population, and to integrate it into a mobile application for use in both clinical and community settings. The study is structured into three phases. Phase 1 involves forward-backward translation of PainPREDICT into Thai, with expert panel review, pilot testing, and psychometric validation. Reliability will be assessed using internal consistency (Cronbach's alpha) and test-retest intraclass correlation coefficients, while validity will be examined through correlations with existing neuropathic pain measures (e.g., DN4) and neurophysiological studies (nerve conduction study, quantitative sensory testing). Phase 2 focuses on the design, development, and usability testing of a mobile application embedding the Thai PainPREDICT questionnaire. Clinicians and patients will test the application, and usability will be assessed with the System Usability Scale and qualitative interviews. Phase 3 evaluates diagnostic accuracy and real-world usability in 200-300 patients with type 1 or type 2 diabetes, including subgroup analysis in resource-limited settings. Diagnostic performance (sensitivity, specificity, positive and negative predictive values, ROC AUC) will be compared with physician diagnosis and objective neurophysiological tests.

Eligible participants are adults (≥18 years) with type 1 or type 2 diabetes who are able to communicate in Thai and provide informed consent. Patients with neuropathy from non-diabetic causes or significant cognitive impairment will be excluded. Recruitment will take place at Chula Neuroscience Center, King Chulalongkorn Memorial Hospital, and affiliated diabetes clinics. The study anticipates enrolling approximately 277 participants, which provides adequate power for psychometric validation and diagnostic accuracy testing. Both PDN patients and diabetic controls without PDN will be included to enable comparative analysis.

The primary outcome is the reliability and validity of the Thai PainPREDICT questionnaire for PDN screening. Secondary outcomes include usability of the mobile application, diagnostic accuracy compared with clinical and neurophysiological standards, and effectiveness in increasing PDN detection in resource-limited settings. The study also seeks to generate evidence on patient and provider satisfaction with the mobile platform. Data will be collected securely, stored in REDCap, and managed in compliance with Thai data protection regulations (PDPA 2019). Ethical approval will be obtained from the Institutional Review Board, Faculty of Medicine, Chulalongkorn University, and written informed consent will be required from all participants.

The expected benefit of this project is the development of a reliable and culturally valid Thai version of PainPREDICT, coupled with an accessible mobile application. This tool is anticipated to facilitate earlier detection of PDN, improve patient management pathways, and reduce disparities in access to care across Thailand. The study will also provide a model for adapting digital health screening tools for other populations with high diabetes burden. Ultimately, the project aims to strengthen evidence-based screening and management of neuropathic pain, improve patient quality of life, and contribute to the broader application of mHealth in chronic disease management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Diagnosed with type 1 diabetes mellitus or type 2 diabetes mellitus.
* Able to communicate in Thai.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Presence of neuropathy due to other causes (e.g., alcohol, chemotherapy, HIV, other systemic diseases).
* Significant cognitive impairment or neurological conditions that prevent comprehension of the questionnaire.
* Severe psychiatric illness that interferes with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-08-27 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Reliability and Validity of Thai PainPREDICT Questionnaire | Baseline through 12 months (Phases 1 and 2)
  Reliability will be assessed by internal consistency (Cronbach's alpha) and test-retest intraclass correlation coefficients. Validity will be examined by correlation with other neuropathic pain questionnaires (DN4, NPSI), construct validity, and diagnostic performance (sensitivity, specificity, ROC AUC) compared with clinical diagnosis and neurophysiological testing.

SECONDARY OUTCOMES:
Usability of the Thai PainPREDICT Mobile Application | Months 7-15 (Phase 2)
  System Usability Scale (SUS) score and qualitative interviews with clinicians and patients to assess ease of use, clarity, efficiency, and satisfaction with the application.
Diagnostic Accuracy of Thai PainPREDICT Questionnaire in Clinical Setting | Months 16-26 (Phase 3)
  Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and ROC AUC of the Thai PainPREDICT questionnaire administered via the mobile application compared with physician diagnosis and neurophysiological tests (NCS, QST).

CONTACTS AND LOCATIONS:
Overall Officials: Jakkrit Amornvit, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- King Chulalongkorn Memorial hospital, The Thai Red Cross Society, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this trial (after de-identification) will be made available to qualified researchers. This includes anonymized questionnaire data, clinical outcome measures, and diagnostic accuracy results. Neurophysiological raw data (e.g., NCS, QST) and laboratory results will also be included in de-identified form. Personal identifiers will be removed to comply with the Thai Personal Data Protection Act (PDPA 2019).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available beginning 12 months after publication of the main results and for up to 5 years thereafter.
Access Criteria: Researchers with a methodologically sound proposal may request access by contacting the principal investigator at Chulalongkorn University. Requests will be reviewed by the study steering committee. Data will be shared through a secure platform with a signed data access agreement.